CLINICAL TRIAL: NCT03888781
Title: Long Term Follow Up and Outcome of Left Ventricular Remodeling in ST Segment Myocardial Infarction Patients After Primary Percutaneous Coronary Intervention
Brief Title: Long Term Follow Up and Outcome of Left Ventricular Remodeling in ST Segment Myocardial Infarction Patients After pPCI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yara Amir Adly Eskander, Principal Investigator, Assiut University
Other Study IDs: Long Term LV Remodeling
Record Dates: First submitted 2019-03-08; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Left Ventricle Remodeling
MeSH Terms: conditions — Ventricular Remodeling | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Left Ventricular Remodeling: By Echocardiography
  Interventions: Device: Echocardiography
- Without Left Ventricular Remodeling: By Echocardiography
  Interventions: Device: Echocardiography

INTERVENTIONS:
Device: Echocardiography — An echocardiogram (also called an echo) is a type of ultrasound test that uses high-pitched sound waves that are sent through a device called a transducer. The device picks up echoes of the sound waves as they bounce off the different parts of your heart. These echoes are turned into moving pictures of your heart that can be seen on a video screen.

SUMMARY:
* To detect long-term effects of left ventricular remodeling in STEMI patients undergoing PPCI.
* And to evaluate outcome.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) with its accompanying adverse sequelae remains one of the most common causes of morbidity and mortality in the world .

Reperfusion therapy is by far the most important therapy for the treatment of acute MI. Reperfusion of the ischemic myocardium reduces the infarct size and improves left ventricular function, both of which contribute to an improved clinical outcome in patients with acute MI .

Using primary PCI has reduced the mortality of patients with acute MI . However, the increased survival rate resulted in the increased incidence of cardio vascular events mainly due to LV remodeling and congestive heart failure .

Post-infarct ventricular remodeling develops in about 30% of patients with a history of myocardial infarction. Ventricular remodeling is a predictor of heart failure and for this reason it assumes a negative prognostic value .

Left ventricular remodeling after ST-segment elevation myocardial infarction (STEMI) treated with primary percutaneous coronary intervention is a major determinant for the short-term and long-term clinical outcomes . Adverse left ventricular remodeling refers to alterations in ventricular architecture involving both the infarcted and non-infarcted zones leading to progressive increase in systolic and diastolic left ventricular volumes.

Left ventricular remodeling following a ST-segment elevated myocardial infarction (STEMI) is an adaptive response to maintain the cardiac output despite myocardial tissue loss. Limited studies have evaluated long term ventricular function after STEMI.

Left Ventricular remodeling, both positive and negative, is an ongoing process and continues at least up to 2 years after STEMI, involving the infarct zone and remote zones. Long-term left ventricular ejection fraction (LVEF) deterioration is characterized by an increase in end-systolic volume and less wall thickening in the remote zones. Patients with long-term LVEF improvement exhibit an increase in left ventricular wall thickening both in the transmural infarct and remote zones. For elucidation of long term effects of left ventricular remodeling, the current study is conducted.

ELIGIBILITY:
Inclusion Criteria:

* All patients were treated successfully by primary PCI more than 2 years ago within 12 hours of onset of chest pain or up to 24 hour of onset of chest pain if there was ongoing ischemia at Assiut University Cardiac Hospital Cath. lab.

Exclusion Criteria:

* Patients with clinical manifestations of acute heart failure or cardiogenic shock at presentation.
* Significant Mitral regurgitation or valve disease.
* Patients with permanent pacemaker insertion.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * It is a cross sectional observational study conducted in Asyut University Cardiac Hospital for STEMI patients to whom PPCI were done. The study includes 127 acute STEMI patients to whom PPCI were done more than 2 years ago.
  * History and clinical examination, ECG diagnosis and location of STEMI, Angiographic study, 2D Echocardiographic examination were done to them.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Long term effect of primary percutaneous coronary intervention on left ventricular remodeling, as measured by change in left ventricular ejection fraction (LVEF) at one year | one year
  Left ventricular remodeling follow up to 127 of acute STEMI patients to whom PPCI were done by 2D Echocardiography measurement to left ventricular ejection fraction change by modified simpthon method

REFERENCES:
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2013 update: a report from the American Heart Association. Circulation. 2013 Jan 1;127(1):e6-e245. doi: 10.1161/CIR.0b013e31828124ad. Epub 2012 Dec 12. No abstract available. PMID 23239837
- [Background] Rossini R, Senni M, Musumeci G, Ferrazzi P, Gavazzi A. Prevention of left ventricular remodelling after acute myocardial infarction: an update. Recent Pat Cardiovasc Drug Discov. 2010 Nov;5(3):196-207. doi: 10.2174/157489010793351999. PMID 20874671
- [Background] Lunde K, Solheim S, Aakhus S, Arnesen H, Abdelnoor M, Egeland T, Endresen K, Ilebekk A, Mangschau A, Fjeld JG, Smith HJ, Taraldsrud E, Grogaard HK, Bjornerheim R, Brekke M, Muller C, Hopp E, Ragnarsson A, Brinchmann JE, Forfang K. Intracoronary injection of mononuclear bone marrow cells in acute myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1199-209. doi: 10.1056/NEJMoa055706. PMID 16990383
- [Background] Flachskampf FA, Schmid M, Rost C, Achenbach S, DeMaria AN, Daniel WG. Cardiac imaging after myocardial infarction. Eur Heart J. 2011 Feb;32(3):272-83. doi: 10.1093/eurheartj/ehq446. Epub 2010 Dec 16. PMID 21163851
- [Background] St John Sutton M, Pfeffer MA, Moye L, Plappert T, Rouleau JL, Lamas G, Rouleau J, Parker JO, Arnold MO, Sussex B, Braunwald E. Cardiovascular death and left ventricular remodeling two years after myocardial infarction: baseline predictors and impact of long-term use of captopril: information from the Survival and Ventricular Enlargement (SAVE) trial. Circulation. 1997 Nov 18;96(10):3294-9. doi: 10.1161/01.cir.96.10.3294. PMID 9396419
- [Background] Opie LH, Commerford PJ, Gersh BJ, Pfeffer MA. Controversies in ventricular remodelling. Lancet. 2006 Jan 28;367(9507):356-67. doi: 10.1016/S0140-6736(06)68074-4. PMID 16443044
- [Background] Cohn JN, Ferrari R, Sharpe N. Cardiac remodeling--concepts and clinical implications: a consensus paper from an international forum on cardiac remodeling. Behalf of an International Forum on Cardiac Remodeling. J Am Coll Cardiol. 2000 Mar 1;35(3):569-82. doi: 10.1016/s0735-1097(99)00630-0. PMID 10716457